CLINICAL TRIAL: NCT05634824
Title: The Combination of IVIg and Low Does Recombinant Human Thrombopoietin for the Management of Immune Thrombocytopenia in Pregnancy
Brief Title: IVIg Plus Low Dose rhTPO for ITP in Pregnancy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiao Hui Zhang, Peking University People's Hospital, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PKU-ITP022
Record Dates: First submitted 2022-11-23; First posted 2022-12-02 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Immune Thrombocytopenia; Pregnancy Related
Keywords: immune thrombocytopenia; pregnancy related
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Immunoglobulins, Intravenous; Thrombopoietin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IVIg plus low dose rhTPO (Experimental): Patients were randomized into experimental and control groups. For the experimental patients, the initial combination therapy consisted rhTPO at an initial does of 150U/kg once daily subcutaneously for 28 days and IVIg 400mg/kg per day for 5 days. If the platelet count was in the range of 30 to 50 × 10^9/L, the combination therapy was repeated. To reduce the risk for thrombocytosis, patients received maintenance therapy consisting rhTPO at a dose of 150U/kg per day if the platelet count rose above 50 × 10^9/L, and treatment discontinued when platelet counts exceeded 100 × 10^9/L. After delivery, the treatment consisted rhTPO 150U/kg per day, and maintained the dose if the platelet count exceeded 30 × 10^9/L. In addition, IVIg 400mg/kg per day for 5 days was added if the platelet count could not maintain above 30 × 10^9/L. If patients did not achieve 30 × 10^9/L within 4 weeks treatment was also discontinued.
  Interventions: Drug: intravenous immunoglobulin plus low dose recombinant human thrombopoietin (rhTPO)
- IvIg treatment (Active Comparator): Patients would be treated with IVIg 400mg/kg per day for 5 days monthly. And treatment discontinued when platelet counts exceeded 100 × 10^9/L.
  Interventions: Drug: intravenous immunoglobulin

INTERVENTIONS:
Drug: intravenous immunoglobulin plus low dose recombinant human thrombopoietin (rhTPO) — rhTPO at an initial does of 150U/kg qd subcutaneously for 28 days and IVIg 400mg/kg qd for 5 days. The maintenance treatment consisted rhTPO 150U/kg qd.
  Arms: IVIg plus low dose rhTPO
Drug: intravenous immunoglobulin — intravenous immunoglobulin
  Arms: IvIg treatment

SUMMARY:
Randomized, open-label, multicenter study to investigate the efficacy and safety of IVIg plus low-dose recombinant thrombopoietin in pregnant patients with corticosteroid or IVIg monotherapy-resistant ITP.

DETAILED DESCRIPTION:
Primary immune thrombocytopenia (ITP) is a common autoimmune disease characterized by a low platelet count resulting from antibody-mediated platelet destruction and insufficient platelet production. ITP, with a prevalence of 1 in 1000-10 000 pregnancies, accounts for about 3% of all causes of thrombocytopenia in pregnancy and is reported to be the most common cause of thrombocytopenia in the first and early second trimesters. It is revealed that severe ITP is associated with devastating outcomes (e.g., postpartum hemorrhage, placental abruption, significant bleeding complication in both women patients and neonates, and even fetal death). It remains a challenge to manage pregnant patients with ITP. First-line treatment options in pregnant ITP patients include corticosteroids and intravenous immunoglobulin (IVIg) currently. However, previous studies reported that the response rate of pregnant ITP patients to corticosteroids was less than 40% and that to IVIg was 38%-56%, which was lower than that of nonpregnant ITP patients. The second-line treatment options are limited for pregnant ITP patients who have no response to the first-line treatments and no agreement has been reached about the optimum second-line treatment for pregnant ITP patients. In addition, single-agent therapy requires an increased dose of the agent and a long-term exposure, which is associated with an increased risk of treatment-related adverse effects. Therefore, the combination of agents sharing disparate mechanisms in the treatment of ITP might be a promising option to maximize efficacy while minimizing side effects.

Thrombopoietin (TPO) mimetics, including eltrombopag and romiplostim, are recommended to be used in the management of nonpregnant corticosteroid-resistant or relapsed ITP patients. However, they may pass through the placenta to have an influence on the fetus, which hinder their use in the management of pregnant ITP patients. Recombinant human thrombopoietin (rhTPO), a full-length and glycosylated TPO with a molecular weight of 90 000 Daltons developed by 3SBIO (Shenyang, China), has also been approved by the China State Food and Drug Administration as a second-line option for nonpregnant ITP patients. It could not cross the placenta theoretically with such a large molecular weight, and thus it has an apparent theoretical advantage over the two TPO mimetics since it would not impact the fetus. Previous data of a multicenter randomized phase 3 clinical trial on nonpregnant ITP patients resistant to corticosteroids showed that rhTPO increased platelet counts rapidly. A study investigating the application of rhTPO in pregnancy suggested rhTPO was a potentially effective and well-tolerated treatment option for ITP patients during pregnancy. A previous case report described a patient with refractory ITP who failed to response to monotherapy of IVIg and TPO mimetics, but responded rapidly with the combination of IVIg and TPO mimetics. It might be explained that the development of ITP was associated with increased platelet destruction and impaired platelet production, and the combination of IVIg and TPO mimetics directed to these two targets since IVIg could reduce platelet destruction whereas TPO mimetics could increase platelet production. Therefore, we conducted a multicenter, single-arm, open-label study to investigate the efficacy and safety of low dose rhTPO plus IVIg in pregnant corticosteroids/IVIg monotherapy-resistant ITP patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients have a diagnosis of primary ITP before or first onset during pregnancy; Patients ≥ 18 years; patients complicate with bleeding manifestations and/or have a platelet count < 30 × 10^9/L and failed to respond to initial treatment of corticosteroids or intravenous immunoglobulin (IVIg) monotherapy or relapsed during the tapering or discontinuation of corticosteroids.

Exclusion Criteria:

* Patients whose thrombocytopenia was secondary to cancer (solid tumor or leukemia), infections, preeclampsia, and HELLP syndrome (hemolysis, elevated liver enzymes, low platelets), and those who had primary immune deficiency, and other hematology or connective tissue diseases during follow-up; patients have heart, kidney, liver, or lung dysfunction; patients received chemotherapy or anticoagulants within 3 months before screening or other second-line ITP-specific treatments within 3 months before screening.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — The study focuses on Pregnancy ITP, the gender of which is female.
Enrollment: 50 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
4-week response rate | 4 weeks

SECONDARY OUTCOMES:
Time to relapse | 13 months
  the interval from response to platelet count of less than 30 × 10^9/L
Bleeding manifestations | 13 months
  presence of bleeding
Additional ITP therapy | 13 months
  Starting of additional ITP therapy
Maternal and neonatal adverse events | 13 months
  According to the Common Terminology Criteria for Adverse Events, Version 6.0
Neonatal platelet count | up to 34 weeks
  at birth, day 7 and day 42